CLINICAL TRIAL: NCT01413854
Title: "Antiinflammatoriska läkemedels Effekt för Att Minska Suicidalitet Hos Deprimerade Patienter Som Nyligen Har Gjort självmordsförsök"
Brief Title: Diclofenac add-on to Treatment as Usual for Suicidal Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not enough recources.
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: eudraCT number 2010-021024-10
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Depression Suicidal
MeSH Terms: interventions — Sugars; Diclofenac; Adrenomedullin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diclofenac (Active Comparator)
  Interventions: Drug: Diclofenac
- sugar pill (Placebo Comparator)
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: sugar pill — One tablet two times daily during four weeks
  Other Names: One tablet two times daily during four weeks
  Arms: sugar pill
Drug: Diclofenac — 50 mg, two times daily (oral adm.) during four weeks
  Other Names: 50 mg, two times daily (oral adm.) during four weeks
  Arms: diclofenac

SUMMARY:
The purpose of this study is to determine whether diclofenac is effective in the treatment of depressed patients with a recent suicide attempt.

DETAILED DESCRIPTION:
The study will start with a feasibility study including treatment of 10 patients with diclofenac.

ELIGIBILITY:
Inclusion Criteria:

* Depressive disorder
* Montgomery Asberg Rating Scale Score more than 20 p.
* Recent suicide attempt (Treated as inpatient due to a recent suicide attempt)
* Informed consent
* Competence to give informed consent

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Serious somatic disease e.g. serious heart, vascular, hepatic, kidney, pulmonary, intestinal, endocrine, haematological or neurological diseases
* Ongoing substance abuse
* Schizophrenia or other psychotic disorders
* Ongoing psychosis
* Risk factors for cardiovascular events
* Ulcer or gastrointestinal bleeding
* Ongoing Electroconvulsive therapy
* Previous allergic reaction to NSAID, acetylsalicylic acid, sulfonamides or the diclofenac or sugar pill content
* Galactose intolerance, lactase deficiency or glucose-galactose malabsorption
* Ongoing treatment with warfarin or other anticoagulants
* Ongoing treatment with ACE inhibitors or angiotensin II antagonists Ongoing treatment with drugs known to effect the immune system Ongoing treatment with rifampicin, carbamazepine or barbiturates

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Suicide Assessment Scale (differences in scores before and after treatment) | four weeks of treatment

SECONDARY OUTCOMES:
Montgomery Asberg Rating Scale (differences in scores before and after treatment) | four weeks of treatment
Barratt Impulsiveness Scale (differences in scores before and after treatment) | four weeks of treatment
Montgomery Asberg depression Ratin scale (changes in suicidality item before and after treatment) | four weeks of treatment
Montgomery Asberg Rating Scale (changes in concentration item before and after treatment) | four weeks of treatment
Comprehensive Psychopathological Rating Scale (changes in aggressive feelings item before and after treatment) | four weeks of treatment
Comprehensive Psychopthological Rating Scale (changes in fatigue item before and after treatment) | four weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Westrin, MD, Phd, Principal Investigator — Lund University
Locations (1):
- Psychiatry Skane, Lund, Sweden